CLINICAL TRIAL: NCT03491215
Title: A Phase I/II Open-label, Single-arm, Multi-center Study of Ruxolitinib Added to Corticosteroids in Pediatric Patients With Grade II-IV Acute Graft vs. Host Disease After Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Study of Pharmacokinetics, Activity and Safety of Ruxolitinib in Pediatric Patients With Grade II-IV Acute Graft vs. Host Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CINC424F12201; 2018-000422-55 (EudraCT Number)
Record Dates: First submitted 2018-03-20; First posted 2018-04-09 (Actual); Results first posted 2024-11-08 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Acute Graft Versus Host Disease
Keywords: Graft versus host disease; GvHD; acute graft versus host disease; aGvHD; Steroid refractory acute graft versus host disease; SR-aGvHD; Ruxolitinib; INC424; allogeneic stem cell transplantation; treatment naive
MeSH Terms: conditions — Graft vs Host Disease | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ruxolitinib (Experimental): All pediatric participants received ruxolitinib twice a day (BID) for a planned duration of 24 weeks in either tablet, capsule or oral solution (liquid), depending on the group they were in.
  Interventions: Drug: Ruxolitinib

INTERVENTIONS:
Drug: Ruxolitinib — All enrolled pediatric participants received ruxolitinib as a 5 mg tablet (adult and adolescent formulation) or an oral pediatric formulation (administered as oral solution or capsule dispersed in liquid).
  Other Names: INC424

SUMMARY:
The study was an open-label, single-arm, Phase I/II multi-center study to investigate the PK, activity and safety of ruxolitinib added to the patient's immunosuppressive regimen in infants, children, and adolescents ages ≥28 days to <18 years old with either grade II-IV aGvHD or grade II-IV SR-aGvHD. The trial design included four age groups: Group 1 included patients ≥12y to <18y, Group 2 included patients ≥6y to <12y, Group 3 included patients ≥2y to <6y, and Group 4 included patients ≥28days to <2y.

DETAILED DESCRIPTION:
This Phase I/II, open-label, uncontrolled, single-arm, multi-center study investigated PK, activity and safety of ruxolitinib when added to the subject's immunosuppressive regimen in infants, children, and adolescents aged ≥ 28 days to < 18 years with either grade II-IV treatment naive acute GvHD or grade II-IV SR-acute GvHD following allogeneic HSCT.

The trial subjects were grouped by age as follows:

* Group 1: subjects ≥ 12y to < 18y,
* Group 2: subjects ≥ 6y to < 12y
* Group 3: subjects ≥ 2y to < 6y
* Group 4 was to include subjects ≥ 28 days to < 2y

Subjects remained in the designated age group throughout the duration of the study, based on their age at the start of treatment. All subjects in this study were enrolled and treated for 24 weeks (approximately 6 months) or until early discontinuation.

All subjects were followed for an additional 18 months (total duration = 2 years from enrolment). Where the occurrence of acute GvHD flare require re-initiation of treatment or when extended tapering resulted in ruxolitinib not having been discontinued by the end of 24 weeks, subjects could continue to taper ruxolitinib beyond 24 weeks up to a maximum of 48 weeks.

Subjects ≥ 12 y to < 18 y (Group 1) were treated with 10 mg BID, this dose was the RP2D, and was used to treat all subjects in this age group in Phase II of Study CINC424F12201. All other age groups were treated with the RP2D determined during Phase I of study CINC424F12201.

Therefore, all ≥12 to <18 year old subjects were automatically enrolled in Phase II. The first 5 subjects treated in Group 1 underwent extensive PK sampling to inform the RP2D determination of the younger age groups in Phase I.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients age ≥28 days and <18 years at the time of informed consent.
* Patients who have undergone alloSCT from any donor source (matched unrelated donor, sibling, haplo-identical) using bone marrow, peripheral blood stem cells, or cord blood. Recipients of myeloablative or reduced intensity conditioning are eligible.
* Patients with a clinically confirmed diagnosis of grades II-IV aGvHD within 48 hours prior to study treatment start. Patients may have either: Treatment-naïve aGvHD (criteria per Harris et al. 2016) OR Steroid refractory aGvHD as per institutional criteria, or per physician decision in case institutional criteria are not available, and the patient is currently receiving systemic corticosteroids.
* Evident myeloid engraftment with ANC > 1,000/µl and platelet count >20,000/µl. (Use of growth factor supplementation and transfusion support is allowed.)

Exclusion Criteria:

* Has received the following systemic therapy for aGvHD: a) Treatment-naïve aGvHD patients have received any prior systemic treatment of aGvHD except for a maximum 72h of prior systemic corticosteroid therapy of methylprednisolone or equivalent after the onset of acute GvHD. Patients are allowed to have received prior GvHD prophylaxis which is not counted as systemic treatment (as long as the prophylaxis was started prior to the diagnosis of aGvHD); OR b) SR-aGvHD patients have received two or more prior systemic treatments for aGvHD in addition to corticosteroids
* Clinical presentation resembling de novo chronic GvHD or GvHD overlap syndrome with both acute and chronic GvHD features (as defined by Jagasia et al 2015).
* Failed prior alloSCT within the past 6 months.
* Presence of relapsed primary malignancy, or who have been treated for relapse after the alloSCT was performed, or who may require rapid immune suppression withdrawal of immune suppression as pre-emergent treatment of early malignancy relapse.
* Acute GvHD occurring after non-scheduled donor leukocyte infusion (DLI) administered for pre-emptive treatment of malignancy recurrence. Note: Patients who have received a scheduled DLI as part of their transplant procedure and not for management of malignancy relapse are eligible.
* Any corticosteroid therapy for indications other than aGvHD at doses > 1 mg/kg/day methylprednisolone (or equivalent prednisone dose 1.25 mg/kg/day) within 7 days of Screening. Routine corticosteroids administered during conditioning or cell infusion is allowed.
* Patients who received JAK inhibitor therapy for any indication after initiation of current alloSCT conditioning.

Other protocol-defined Inclusion/Exclusion may apply.

Ages: 28 Days to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2019-02-21 (Actual); Primary Completion 2021-03-11 (Actual); Study Completion 2023-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (17):
- Belgium (2):
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Laken
- Novartis Investigative Site, Montreal, Quebec, Canada
- Novartis Investigative Site, Copenhagen, Denmark
- France (5):
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Rennes
  - Novartis Investigative Site, Vandœuvre-lès-Nancy
- Italy (2):
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Roma, RM
- Japan (2):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Saitama
- Novartis Investigative Site, Seoul, South Korea
- Spain (3):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent expert panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data is currently available according to the process described on www.clinicalstudydatarequest.com.
URL: http://www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Locatelli F, Kang HJ, Bruno B, Gandemer V, Rialland F, Faraci M, Takahashi Y, Koh K, Bittencourt H, Cleary G, Rosko C, Li X, St Pierre A, Prahallad A, Diaz-de-Heredia C. Ruxolitinib for pediatric patients with treatment-naive and steroid-refractory acute graft-versus-host disease: the REACH4 study. Blood. 2024 Nov 14;144(20):2095-2106. doi: 10.1182/blood.2023022565. PMID 39046767
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1936

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 45 subjects were enrolled in the study and treated with the confirmed RP2D, of which at least 20% had treatment naïve acute GvHD and at least 40% had SR-acute GvHD. The study was a single arm study with the subjects grouped as follows: Group 1: subjects ≥ 12y to < 18y, Group 2: subjects ≥ 6y to < 12y, Group 3: subjects ≥ 2y to < 6y, Group 4 was to include subjects ≥ 28 days to < 2y.
Pre-assignment Details: Five subjects were to be enrolled to each age group with no minimum for Group 4, although no subjects were enrolled in Group 4.
  All subjects participating in Phase I also participated in Phase II so the number of subjects in each phase is identical.
  The study was conducted in 8 countries and 19 centers.
Groups:
- Group 1: Subjects ≥ 12y to < 18y - RUX 10mg BID: All pediatric participants received ruxolitinib (RUX) 10 mg BID
- Group 2: Subjects ≥ 6y to < 12y - RUX 5mg BID: All pediatric participants received RUX 5mg BID.
- Group 3: Subjects ≥ 2y to < 6y - RUX 4mg/m^2 BID: All pediatric participants received RUX 4mg/m^2 BID.
- Group 4: Subjects >= 28 Days to < 2y: Recommend phase 2 dose (RP2D) not defined.
Period: Overall Study
Arm/Group | Group 1: Subjects ≥ 12y to < 18y - RUX 10mg BID | Group 2: Subjects ≥ 6y to < 12y - RUX 5mg BID | Group 3: Subjects ≥ 2y to < 6y - RUX 4mg/m^2 BID | Group 4: Subjects >= 28 Days to < 2y
Started | 18 | 12 | 15 | 0
Rux Formulation - Received Tablet | 18 | 10 | 0 | 0
Rux Formulation - Received Capsule | 0 | 2 | 7 | 0
Rux Formulation - Received Oral Solution | 0 | 0 | 8 | 0
Completed | 11 | 10 | 14 | 0
Not Completed | 7 | 2 | 1 | 0
Not completed — Death | 6 | 2 | 1 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) comprised all subjects to whom study treatment was assigned and who received at least one dose of study treatment. No subjects were enrolled in Group 4.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Subjects ≥ 12y to < 18y - RUX 10mg BID | Group 2: Subjects ≥ 6y to < 12y - RUX 5mg BID | Group 3: Subjects ≥ 2y to < 6y - RUX 4mg/m^2 BID | Group 4: Subjects >= 28 Days to < 2y | Total
Number analyzed (Participants) | 18 | 12 | 15 | 0 | 45
Age, Continuous [Mean (Standard Deviation); unit: Months] | 172.7 (18.94) | 86.1 (11.08) | 45.5 (14.57) |  | 107.2 (58.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 5 | 0 | 17
  Male | 13 | 5 | 10 | 0 | 28
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 11 | 5 | 4 |  | 20
  Asian | 3 | 3 | 5 |  | 11
  Missing -Note: race is not collected in France | 4 | 4 | 6 |  | 14

OUTCOME MEASURES:

1. Primary Outcome: Phase I: Measurement of Pharmacokinetic (PK) Parameter, AUClast, in aGvHD and SR-aGvHD Patients
Description: Measurement in acute GvHD and SR-acute GvHD subjects used extensive PK sampling in Groups 1-3 sparse sampling in Group 4.
  AUClast: The AUC from time zero to the last measurable concentration sampling time (Tlast).
Time Frame: Day 1: at predose, 0.5,1,1.5, 2, 4, 6, 9 hours post dose
Population: PAS: The Pharmacokinetic Analysis Set (PAS) included all subjects who provided at least one evaluable PK concentration. For a concentration to be evaluable, subjects were required to:
  * Take the dose of ruxolitinib prior to PK sample.
  * For pre-dose samples, to not vomit within 2 hours after the previous dosing of ruxolitinib prior to sampling; for post-dose samples, to not vomit within 2 hours after the dosing of ruxolitinib.
  No subjects were enrolled in Group 4.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Groups:
- Group 1: Subjects ≥ 12y to < 18y - RUX 10mg BID Tablet: All pediatric participants received ruxolitinib (RUX) 10 mg BID tablet.
- Group 2: Subjects ≥ 6y to < 12y - RUX 5mg BID Tablet: All pediatric participants received RUX 5mg BID tablet.
- Group 2: Subjects ≥ 6y to < 12y - RUX 5mg BID Capsule: All pediatric participants received RUX 5mg BID capsule.
- Group 3: Subjects ≥ 2y to < 6y - RUX 4mg/m^2 BID Capsule: All pediatric participants received RUX 4mg/m^2 BID capsule.
- Group 3: Subjects ≥ 2y to < 6y - RUX 4mg/m^2 BID Liquid: All pediatric participants received RUX 4mg/m^2 BID liquid.
Arm/Group | Group 1: Subjects ≥ 12y to < 18y - RUX 10mg BID Tablet | Group 2: Subjects ≥ 6y to < 12y - RUX 5mg BID Tablet | Group 2: Subjects ≥ 6y to < 12y - RUX 5mg BID Capsule | Group 3: Subjects ≥ 2y to < 6y - RUX 4mg/m^2 BID Capsule | Group 3: Subjects ≥ 2y to < 6y - RUX 4mg/m^2 BID Liquid | Group 4: Subjects >= 28 Days to < 2y
Number analyzed (Participants) | 5 | 8 | 2 | 7 | 8 | 0
ng*hr/mL | 252 (186.6) | 372 (58.6) | 154 (58.1) | 239 (65.3) | 259 (53.6) |
Statistical Analysis 1: Comparison: Group 2: Subjects ≥ 6y to < 12y - RUX 5mg BID Tablet vs Group 2: Subjects ≥ 6y to < 12y - RUX 5mg BID Capsule vs Group 3: Subjects ≥ 2y to < 6y - RUX 4mg/m^2 BID Capsule vs Group 3: Subjects ≥ 2y to < 6y - RUX 4mg/m^2 BID Liquid; Group 3 vs Group 2; Test type: Other — Comparison; GMR = 0.801, 90% CI 2-sided [0.490 to 1.311]
Statistical Analysis 2: Comparison: Group 1: Subjects ≥ 12y to < 18y - RUX 10mg BID Tablet vs Group 3: Subjects ≥ 2y to < 6y - RUX 4mg/m^2 BID Capsule vs Group 3: Subjects ≥ 2y to < 6y - RUX 4mg/m^2 BID Liquid; Group 3 vs. Group 1; Test type: Other — Comparison; GMR = 0.991, 90% CI 2-sided [0.532 to 1.846]
Statistical Analysis 3: Comparison: Group 1: Subjects ≥ 12y to < 18y - RUX 10mg BID Tablet vs Group 2: Subjects ≥ 6y to < 12y - RUX 5mg BID Tablet vs Group 2: Subjects ≥ 6y to < 12y - RUX 5mg BID Capsule; Group 2 vs. Group 1; Test type: Other — Comparison; GMR = 1.237, 90% CI 2-sided [0.639 to 2.394]

2. Primary Outcome: Phase I: Measurement of PK Parameter, Cmax, in aGvHD and SR-aGvHD Patients
Description: Measurement in acute GvHD and SR-acute GvHD subjects used extensive PK sampling in Groups 1-3 and sparse sampling in Group 4.
  Cmax: The maximum (peak) observed plasma drug concentration
Time Frame: Day 1: at predose, 0.5,1,1.5, 2, 4, 6, 9 hours post dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/ML
Arm/Group | Group 1: Subjects ≥ 12y to < 18y - RUX 10mg BID Tablet | Group 2: Subjects ≥ 6y to < 12y - RUX 5mg BID Tablet | Group 2: Subjects ≥ 6y to < 12y - RUX 5mg BID Capsule | Group 3: Subjects ≥ 2y to < 6y - RUX 4mg/m^2 BID Capsule | Group 3: Subjects ≥ 2y to < 6y - RUX 4mg/m^2 BID Liquid | Group 4: Subjects >= 28 Days to < 2y
Number analyzed (Participants) | 5 | 8 | 2 | 7 | 8 | 0
ng/ML | 66.1 (169.8) | 105 (71.4) | 49.4 (45.7) | 61.2 (81.1) | 66.5 (60.8) |
Statistical Analysis 1: Comparison: Group 2: Subjects ≥ 6y to < 12y - RUX 5mg BID Tablet vs Group 2: Subjects ≥ 6y to < 12y - RUX 5mg BID Capsule vs Group 3: Subjects ≥ 2y to < 6y - RUX 4mg/m^2 BID Capsule vs Group 3: Subjects ≥ 2y to < 6y - RUX 4mg/m^2 BID Liquid; Group 3 vs. Group 2; Test type: Other — Comparison; GMR = 0.709, 90% CI 2-sided [0.425 to 1.184]
Statistical Analysis 2: Comparison: Group 1: Subjects ≥ 12y to < 18y - RUX 10mg BID Tablet vs Group 3: Subjects ≥ 2y to < 6y - RUX 4mg/m^2 BID Capsule vs Group 3: Subjects ≥ 2y to < 6y - RUX 4mg/m^2 BID Liquid; Group 3 vs. Group 1; Test type: Other — Comparison; GMR = 0.968, 90% CI 2-sided [0.506 to 1.851]
Statistical Analysis 3: Comparison: Group 1: Subjects ≥ 12y to < 18y - RUX 10mg BID Tablet vs Group 2: Subjects ≥ 6y to < 12y - RUX 5mg BID Tablet vs Group 2: Subjects ≥ 6y to < 12y - RUX 5mg BID Capsule; Group 2 vs. Group 1; Test type: Other — Comparison; GMR = 1.365, 90% CI 2-sided [0.686 to 2.714]

3. Primary Outcome: Phase I: Measurement of PK Parameter, T1/2, in aGvHD and SR-aGvHD Patients
Description: Measurement in acute GvHD and SR-acute GvHD subjects used extensive PK sampling in Groups 1-3 and sparse sampling in Group 4.
  T1/2: The elimination half-life associated with the terminal slope (Lambda_z ) of a semi logarithmic concentration-time curve
Time Frame: Day 1: at predose, 0.5,1,1.5, 2, 4, 6, 9 hours post dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | Group 1: Subjects ≥ 12y to < 18y - RUX 10mg BID Tablet | Group 2: Subjects ≥ 6y to < 12y - RUX 5mg BID Tablet | Group 2: Subjects ≥ 6y to < 12y - RUX 5mg BID Capsule | Group 3: Subjects ≥ 2y to < 6y - RUX 4mg/m^2 BID Capsule | Group 3: Subjects ≥ 2y to < 6y - RUX 4mg/m^2 BID Liquid | Group 4: Subjects >= 28 Days to < 2y
Number analyzed (Participants) | 2 | 5 | 2 | 5 | 5 | 0
hour | 1.33 (31.7) | 1.66 (17.5) | 1.50 (6.5) | 1.86 (29.9) | 1.78 (66.3) |

4. Primary Outcome: Phase I: Measurement of PK Parameter, Ctrough, in aGvHD and SR-aGvHD Patients
Description: Measurement in acute GvHD and SR-acute GvHD subjects used extensive PK sampling in Groups 1-3 and sparse sampling in Group 4. Ctrough: The minimum observed plasma concentration at the end of an administration interval (corresponding to the pre-dose concentration prior to the following administration).
Time Frame: Day 7 at pre-dose
Population: PAS: The Pharmacokinetic Analysis Set (PAS) included all subjects who provided at least one evaluable PK concentration. For a concentration to be evaluable, subjects were required to:
  * Take the dose of ruxolitinib prior to PK sample.
  * For pre-dose samples, not vomit within 2 hours after the previous dosing of ruxolitinib prior to sampling; for post-dose samples, to not vomit within 2 hours after the dosing of ruxolitinib.
  No subjects were enrolled in Group 4.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/ml
Arm/Group | Group 1: Subjects ≥ 12y to < 18y - RUX 10mg BID Tablet | Group 2: Subjects ≥ 6y to < 12y - RUX 5mg BID Tablet | Group 2: Subjects ≥ 6y to < 12y - RUX 5mg BID Capsule | Group 3: Subjects ≥ 2y to < 6y - RUX 4mg/m^2 BID Capsule | Group 3: Subjects ≥ 2y to < 6y - RUX 4mg/m^2 BID Liquid | Group 4: Subjects >= 28 Days to < 2y
Number analyzed (Participants) | 7 | 6 | 2 | 6 | 8 | 0
ng/ml | 9.27 (379.4) | 9.75 (255.5) | 1.71 (1.2) | 6.18 (195.8) | 3.99 (277.1) |
Statistical Analysis 1: Comparison: Group 2: Subjects ≥ 6y to < 12y - RUX 5mg BID Tablet vs Group 2: Subjects ≥ 6y to < 12y - RUX 5mg BID Capsule vs Group 3: Subjects ≥ 2y to < 6y - RUX 4mg/m^2 BID Capsule vs Group 3: Subjects ≥ 2y to < 6y - RUX 4mg/m^2 BID Liquid; Group 3 vs. Group 2; Test type: Other — Comparison; GMR = 0.759, 90% CI 2-sided [0.245 to 2.352]
Statistical Analysis 2: Comparison: Group 1: Subjects ≥ 12y to < 18y - RUX 10mg BID Tablet vs Group 3: Subjects ≥ 2y to < 6y - RUX 4mg/m^2 BID Capsule vs Group 3: Subjects ≥ 2y to < 6y - RUX 4mg/m^2 BID Liquid; Group 3 vs. Group 1; Test type: Other — Comparison; GMR = 0.516, 90% CI 2-sided [0.150 to 1.784]
Statistical Analysis 3: Comparison: Group 1: Subjects ≥ 12y to < 18y - RUX 10mg BID Tablet vs Group 2: Subjects ≥ 6y to < 12y - RUX 5mg BID Tablet vs Group 2: Subjects ≥ 6y to < 12y - RUX 5mg BID Capsule; Group 2 vs. Group 1; Test type: Other — Comparison; GMR = 0.681, 90% CI 2-sided [0.178 to 2.597]

5. Primary Outcome: Phase I: Age-based Determination of Recommended Phase 2 Dose (RP2D) Using AUClast
Description: Phase I: Age-based determination of RP2D in Groups 2 and 3 and was based on observed PK parameters in Groups 1-3
  * Group 2: age ≥ 6 to < 12 years
  * Group 3: age ≥ 2 to < 6 years AUClast: The AUC from time zero to the last measurable concentration sampling time (Tlast).
Time Frame: Day 1: at predose, 0.5,1,1.5, 2, 4, 6, 9 hours post dose
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Groups:
- Group 2: Subjects ≥ 6y to < 12y - RUX 5mg BID Tablet: All patients received RUX 5mg BID tablet in addition to corticosteroids +/-calcineurin inhibitor (CNI)
- Group 3: Subjects ≥ 2y to < 6y - RUX 4mg/m^2 BID Capsule: All patients received RUX 4mg/m^2 BID capsule in addition to corticosteroids +/- calcineurin inhibitor (CNI)
- Group 3: Subjects ≥ 2y to < 6y - RUX 4mg/m^2 BID Liquid: All patients received RUX 4mg/m^2 BID liquid in addition to corticosteroids +/-calcineurin inhibitor (CNI)
Arm/Group | Group 1: Subjects ≥ 12y to < 18y - RUX 10mg BID Tablet | Group 2: Subjects ≥ 6y to < 12y - RUX 5mg BID Capsule | Group 2: Subjects ≥ 6y to < 12y - RUX 5mg BID Tablet | Group 3: Subjects ≥ 2y to < 6y - RUX 4mg/m^2 BID Capsule | Group 3: Subjects ≥ 2y to < 6y - RUX 4mg/m^2 BID Liquid | Group 4: Subjects >= 28 Days to < 2y
Number analyzed (Participants) | 5 | 2 | 8 | 7 | 8 | 0
h*ng/mL | 252 (186.6) | 154 (58.1) | 372 (58.6) | 239 (65.3) | 259 (53.6) |

6. Primary Outcome: Phase I: Age-based Determination of Recommended Phase 2 Dose (RP2D) Using Cmax
Description: Phase I: Age-based determination of RP2D in Groups 2 and 3 and was based on observed PK parameters in Groups 1-3
  * Group 2: age ≥ 6 to < 12 years
  * Group 3: age ≥ 2 to < 6 years Cmax: The maximum (peak) observed plasma drug concentration.
Time Frame: Day 1: at predose, 0.5,1,1.5, 2, 4, 6, 9 hours post dose
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Group 1: Subjects ≥ 12y to < 18y - RUX 10mg BID Tablet | Group 2: Subjects ≥ 6y to < 12y - RUX 5mg BID Capsule | Group 2: Subjects ≥ 6y to < 12y - RUX 5mg BID Tablet | Group 3: Subjects ≥ 2y to < 6y - RUX 4mg/m^2 BID Capsule | Group 3: Subjects ≥ 2y to < 6y - RUX 4mg/m^2 BID Liquid | Group 4: Subjects >= 28 Days to < 2y
Number analyzed (Participants) | 5 | 2 | 8 | 7 | 8 | 0
ng/mL | 66.1 (169.8) | 49.4 (45.7) | 105 (71.4) | 61.2 (81.1) | 66.5 (60.8) |

7. Primary Outcome: Phase I: Age-based Determination of Recommended Phase 2 Dose (RP2D) Using Ctrough
Description: Phase I: Age-based determination of RP2D in Groups 2 and 3 and was based on observed PK parameters in Groups 1-3
  * Group 2: age ≥ 6 to < 12 years
  * Group 3: age ≥ 2 to < 6 years Ctrough: The minimum observed plasma concentration at the end of an administration interval (corresponding to the pre-dose concentration prior to the following administration).
Time Frame: Day 7 at pre-dose
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/ml
Arm/Group | Group 1: Subjects ≥ 12y to < 18y - RUX 10mg BID Tablet | Group 2: Subjects ≥ 6y to < 12y - RUX 5mg BID Capsule | Group 2: Subjects ≥ 6y to < 12y - RUX 5mg BID Tablet | Group 3: Subjects ≥ 2y to < 6y - RUX 4mg/m^2 BID Capsule | Group 3: Subjects ≥ 2y to < 6y - RUX 4mg/m^2 BID Liquid | Group 4: Subjects >= 28 Days to < 2y
Number analyzed (Participants) | 6 | 2 | 8 | 6 | 8 | 0
ng/ml | 8.85 (538.6) | 1.71 (1.2) | 10.6 (208.1) | 6.18 (195.8) | 3.99 (277.1) |

8. Primary Outcome: Phase II: Overall Response Rate (ORR)
Description: Phase II: ORR is defined as the percentage of patients demonstrating a complete response (CR) or partial response (PR) without requirement for additional systemic therapies for an earlier progression, mixed response or non-response. Scoring of response was relative to the organ stage at the start of the study treatment.
  Complete response (CR) is defined as a score of 0 for the aGvHD grading in all evaluable organs that indicates complete resolution of all signs and symptoms of aGvHD in all evaluable organs without administration of additional systemic therapy for any earlier progression, mixed response or non-response of aGvHD.
  Partial response (PR) is defined as improvement of 1 stage in 1 or more organs involved with aGvHD signs or symptoms without progression in other organs or sites without administration of additional systemic therapy for an earlier progression, mixed response or non-response of aGvHD.
Time Frame: Day 28
Population: The Efficacy Evaluable Set (EES) comprised all subjects to whom study treatment was assigned at the recommended phase 2 dose (RP2D) of ruxolitinib and who received at least one dose of study treatment at that dose level. No subjects were enrolled in Group 4.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: Subjects ≥ 12y to < 18y - RUX 10mg BID | Group 2: Subjects ≥ 6y to < 12y - RUX 5mg BID | Group 3: Subjects ≥ 2y to < 6y - RUX 4mg/m^2 BID | Group 4: Subjects >= 28 Days to < 2y
Number analyzed (Participants) | 18 | 12 | 15 | 0
Percentage of participants | 83.3 [62.3 to 95.3] | 83.3 [56.2 to 97.0] | 86.7 [63.7 to 97.6] |

9. Secondary Outcome: Percentage of All Patients Who Achieved a Complete Response (CR) or Partial Response (PR) (Durable Overall Response Rate (ORR))
Description: Durable ORR at Day 56 was defined as the percentage of all subjects who achieved a complete response (CR) or partial response (PR) at Day 28 and maintained a CR or PR at Day 56.
  Complete-response was defined as a score of 0 for the acute GvHD grading in all evaluable organs that indicates complete resolution of all signs and symptoms of acute GvHD in all evaluable organs without administration of additional systemic therapies for any earlier progression, mixed response or non-response of acute GvHD.
  Partial response was defined as improvement of 1 stage in 1 or more organs involved with acute GvHD signs or symptoms without progression in other organs or sites without administration of additional systemic therapies for an earlier progression, mixed response or non-response of acute GvHD.
Time Frame: Day 56
Population: The Efficacy Evaluable Set (EES) comprised all subjects to whom study treatment was assigned at the RP2D of ruxolitinib and who received at least one dose of study treatment at that dose level. No subjects were enrolled in Group 4.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: Subjects ≥ 12y to < 18y - RUX 10mg BID | Group 2: Subjects ≥ 6y to < 12y - RUX 5mg BID | Group 3: Subjects ≥ 2y to < 6y - RUX 4mg/m^2 BID | Group 4: Subjects >= 28 Days to < 2y
Number analyzed (Participants) | 18 | 12 | 15 | 0
Percentage of participants | 55.6 [34.1 to 75.6] | 75.0 [47.3 to 92.8] | 73.3 [48.9 to 90.3] |

10. Secondary Outcome: Percentage of Patients Who Achieved OR (CR+PR) at Day 14
Description: ORR at Day 14 was defined as the percentage of participants with complete response (CR) or partial response (PR ) at Day 14 according to standard criteria.
  Complete response (CR) is defined as a score of 0 for the aGvHD grading in all evaluable organs that indicates complete resolution of all signs and symptoms of aGvHD in all evaluable organs without administration of additional systemic therapy for any earlier progression, mixed response or non-response of aGvHD.
  Partial response (PR) is defined as improvement of 1 stage in 1 or more organs involved with aGvHD signs or symptoms without progression in other organs or sites without administration of additional systemic therapy for an earlier progression, mixed response or non-response of aGvHD.
Time Frame: Day 14
Population: as for outcome 9
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: Subjects ≥ 12y to < 18y - RUX 10mg BID | Group 2: Subjects ≥ 6y to < 12y - RUX 5mg BID | Group 3: Subjects ≥ 2y to < 6y - RUX 4mg/m^2 BID | Group 4: Subjects >= 28 Days to < 2y
Number analyzed (Participants) | 18 | 12 | 15 | 0
Percentage of participants | 72.2 [50.2 to 88.4] | 66.7 [39.1 to 87.7] | 86.7 [63.7 to 97.6] |

11. Secondary Outcome: Area Under the Curve (AUClast) Versus Efficacy: Impact of AUClast on Overall Response Rate (ORR) at Day 28
Description: To assess pharmacokinetic/pharmacodynamic relationship (comparison of AUClast with ORR at day 28). ORR is the percentage of patients with a complete response (CR) or partial response (PR) without additional systemic therapies. Given age group did not have a significant effect on the model fit, the comparison is made indirectly through the odds ratio across exposure levels in each group. A high response rate may prevent model convergence. Results are shown only upon successful convergence.
Time Frame: Day 28
Population: PK-Efficacy set includes 40 subjects from F12201. CR is a score of 0 for the aGvHD grading in all evaluable organs that indicate complete resolution of all signs of aGvHD in all evaluable organs without administration of additional systemic therapy for aGvHD.
  PR is improvement of 1 stage in 1 or more organs involved with aGvHD signs without progression in other organs or sites without administration of additional systemic therapy of aGvHD. No subjects were enrolled in Group 4.
Measure: Number; unit: Percentage of participants
Groups:
- Group 1: Subjects ≥ 12y to < 18y - RUX 10mg BID Tablet: All pediatric participants received ruxolitinib (RUX) 10 mg BID.
Arm/Group | Group 1: Subjects ≥ 12y to < 18y - RUX 10mg BID Tablet | Group 2: Subjects ≥ 6y to < 12y - RUX 5mg BID | Group 3: Subjects ≥ 2y to < 6y - RUX 4mg/m^2 BID | Group 4: Subjects >= 28 Days to < 2y
Number analyzed (Participants) | 14 | 11 | 15 | 0
Percentage of participants | 92.9 | 90.9 | 86.7 |

12. Secondary Outcome: Area Under the Curve (AUClast) Versus Efficacy: Impact of AUClast on Durable Response Rate (DRR) at Day 56
Description: To assess pharmacokinetic/pharmacodynamic relationship (comparison of AUClast with DRR at day 56). Durable ORR at Day 56 was defined as the percentage of all participants who achieved a complete response (CR) or partial response (PR) at Day 28 and maintained a CR or PR at Day 56. Given age group did not have a significant effect on the model fit, the comparison is made indirectly through the odds ratio across exposure levels in each group. A high response rate may prevent model convergence. Results are shown only upon successful convergence.
Time Frame: Day 56
Population: as for outcome 11
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1: Subjects ≥ 12y to < 18y - RUX 10mg BID | Group 2: Subjects ≥ 6y to < 12y - RUX 5mg BID | Group 3: Subjects ≥ 2y to < 6y - RUX 4mg/m^2 BID | Group 4: Subjects >= 28 Days to < 2y
Number analyzed (Participants) | 14 | 11 | 15 | 0
Percentage of participants | 71.4 | 81.8 | 73.3 |
Statistical Analysis 1: Comparison: Group 1: Subjects ≥ 12y to < 18y - RUX 10mg BID vs Group 2: Subjects ≥ 6y to < 12y - RUX 5mg BID; Test type: Superiority; Odds Ratio (OR) = 0.976, 95% CI 2-sided [0.858 to 1.109]
Statistical Analysis 2: Comparison: Group 1: Subjects ≥ 12y to < 18y - RUX 10mg BID vs Group 3: Subjects ≥ 2y to < 6y - RUX 4mg/m^2 BID; Test type: Superiority; Odds Ratio (OR) = 0.951, 95% CI 2-sided [0.735 to 1.232]

13. Secondary Outcome: Area Under the Curve (AUClast) Versus Safety: Impact of AUClast on Bleeding
Description: To assess pharmacokinetic/pharmacodynamic relationship (comparison of AUClast with safety - bleeding). Bleeding was reported as an adverse event and the AE severity grade was assessed according to CTCAE grading. Given age group did not have a significant effect on the model fit, the comparison is made indirectly through the hazard ratio across exposure levels in each group. A high response rate may prevent model convergence. Results are shown only upon successful convergence.
Time Frame: 24 weeks
Population: PK-Safety set includes 40 subjects from F12201. No subjects were enrolled in Group 4.
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1: Subjects ≥ 12y to < 18y - RUX 10mg BID | Group 2: Subjects ≥ 6y to < 12y - RUX 5mg BID | Group 3: Subjects ≥ 2y to < 6y - RUX 4mg/m^2 BID | Group 4: Subjects >= 28 Days to < 2y
Number analyzed (Participants) | 14 | 11 | 15 | 0
Percentage of participants | 21.4 | 18.2 | 6.7 |
Statistical Analysis 1: Comparison: Group 1: Subjects ≥ 12y to < 18y - RUX 10mg BID vs Group 2: Subjects ≥ 6y to < 12y - RUX 5mg BID; Test type: Superiority; Hazard Ratio (HR) = 1.014, 95% CI 2-sided [0.921 to 1.115]
Statistical Analysis 2: Comparison: Group 1: Subjects ≥ 12y to < 18y - RUX 10mg BID vs Group 3: Subjects ≥ 2y to < 6y - RUX 4mg/m^2 BID; Test type: Superiority; Hazard Ratio (HR) = 1.029, 95% CI 2-sided [0.841 to 1.258]

14. Secondary Outcome: Area Under the Curve (AUClast) Versus Safety: Impact of AUClast on Infection
Description: To assess pharmacokinetic/pharmacodynamic relationship (comparison of AUClast with safety - infection). This analysis includes subjects from F12201 (pediatric and adolescent participants) study. Infections were reported as adverse events and the AE severity grade was assessed according to CTCAE grading. Given age group did not have a significant effect on the model fit, the comparison is made indirectly throughs the hazard ratio across exposure levels in each group. A high response rate may prevent model convergence. Results are shown only upon successful convergence
Time Frame: 24 weeks
Population: PK-Safety set includes 40 subjects from F12201. No subjects were enrolled in Group 4.
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1: Subjects ≥ 12y to < 18y - RUX 10mg BID | Group 2: Subjects ≥ 6y to < 12y - RUX 5mg BID | Group 3: Subjects ≥ 2y to < 6y - RUX 4mg/m^2 BID | Group 4: Subjects >= 28 Days to < 2y
Number analyzed (Participants) | 14 | 11 | 15 | 0
Percentage of participants | 64.3 | 63.6 | 60.0 |
Statistical Analysis 1: Comparison: Group 1: Subjects ≥ 12y to < 18y - RUX 10mg BID vs Group 2: Subjects ≥ 6y to < 12y - RUX 5mg BID; Test type: Superiority; Hazard Ratio (HR) = 1.063, 95% CI 2-sided [1.012 to 1.117]
Statistical Analysis 2: Comparison: Group 1: Subjects ≥ 12y to < 18y - RUX 10mg BID vs Group 3: Subjects ≥ 2y to < 6y - RUX 4mg/m^2 BID; Test type: Superiority; Hazard Ratio (HR) = 1.132, 95% CI 2-sided [1.025 to 1.25]

15. Secondary Outcome: Duration of Response (DOR)
Description: Duration of response was defined as the time from first response (PR or CR) until acute GvHD progression, or the date of additional systemic therapy for acute GvHD. Death without prior observation of acute GvHD progression, and onset of chronic GvHD are considered to be competing risks. Duration of response will be censored at the last response assessment prior to or at the analysis cut-off date, if no events/competing risks occurred on or before 4 weeks (28 days) after the last GvHD assessment. The estimated probability of loss of response at 1, 2 and 6 months after participant's first achievement of CR or PR has been reported. Due to the presence of competing risk, the DOR results are being presented in the form of the probability of loss of response at different time points. As planned in the Statistical Analysis Plan (SAP), this outcome measure is provided for all subjects instead of per age groups.
Time Frame: Months 1, 2 & 6
Population: The Efficacy Evaluable Set (EES) comprised all subjects to whom study treatment was assigned at the RP2D of ruxolitinib and who received at least one dose of study treatment at that dose level. The DOR was assessed only for responders (i.e. those with CR or PR) at Day 28. No subjects were enrolled in Group 4.
Measure: Number (95% Confidence Interval); unit: Prob. of loss of response in percentage
Groups:
- All Subjects (Group 1, Group 2 & Group 3): All pediatric participants received ruxolitinib (RUX) regardless of dose and age group.
Arm/Group | All Subjects (Group 1, Group 2 & Group 3) | Group 4: Subjects >= 28 Days to < 2y
Number analyzed (Participants) | 38 | 0
Prob. of loss of response in percentage
  1 Month | 2.63 [0.20 to 11.98] |
  2 Months | 5.41 [0.95 to 16.13] |
  6 Months | 20.37 [8.74 to 35.40] |

16. Secondary Outcome: Weekly Cumulative Steroid Dose for Each Patient up to Day 56
Description: The weekly cumulative steroid dose was calculated for each subject up to Day 56 and the overall cumulative steroid dose was calculated for each subject at Day 56.
Time Frame: up to 56 days (Week 1 - Week 8)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mg/kg
Arm/Group | Group 1: Subjects ≥ 12y to < 18y - RUX 10mg BID | Group 2: Subjects ≥ 6y to < 12y - RUX 5mg BID | Group 3: Subjects ≥ 2y to < 6y - RUX 4mg/m^2 BID | Group 4: Subjects >= 28 Days to < 2y
Number analyzed (Participants) | 18 | 12 | 15 | 0
mg/kg
  Week 1 | 12.6 (6.04) | 14.1 (4.60) | 11.9 (5.32) |
  Week 2 | 21.9 (10.79) | 26.1 (9.91) | 21.0 (8.03) |
  Week 3: number analyzed (Participants) | 17 | 12 | 15 | 0
  Week 3 | 30.1 (16.14) | 36.5 (17.18) | 29.0 (10.20) |
  Week 4: number analyzed (Participants) | 16 | 10 | 14 | 0
  Week 4 | 37.5 (21.19) | 46.9 (24.91) | 36.8 (12.95) |
  Week 5: number analyzed (Participants) | 16 | 10 | 14 | 0
  Week 5 | 42.6 (24.05) | 55.2 (31.52) | 42.0 (14.76) |
  Week 6: number analyzed (Participants) | 13 | 10 | 10 | 0
  Week 6 | 48.9 (24.57) | 61.8 (35.80) | 48.8 (17.68) |
  Week 7: number analyzed (Participants) | 11 | 9 | 10 | 0
  Week 7 | 51.5 (28.34) | 60.6 (35.75) | 53.7 (19.32) |
  Week 8: number analyzed (Participants) | 9 | 7 | 10 | 0
  Week 8 | 61.3 (30.29) | 73.6 (43.11) | 58.1 (20.50) |

17. Secondary Outcome: Overall Survival (OS) Per Kaplan Meier
Description: OS is defined as the time from the start of treatment to the date of death due to any cause. If a subject was not known to have died, then OS was censored at the latest date the subject was known to be alive. The estimated survival probability at 1,2,6,12,18 months after start of treatment has been reported. (on or before the cut-off date). As planned in the SAP, this outcome measure is provided for all subjects instead of per age groups.
Time Frame: 1 Month (M), 2 M, 6M, 12M, 18M
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: survival probability in percentage
Arm/Group | All Subjects (Group 1, Group 2 & Group 3) | Group 4: Subjects >= 28 Days to < 2y
Number analyzed (Participants) | 45 | 0
survival probability in percentage
  1 Month | 100 [100 to 100] |
  2 Months | 100 [100 to 100] |
  6 Months | 93.33 [80.74 to 97.80] |
  12 Months | 88.83 [75.22 to 95.19] |
  18 Months | 79.72 [64.64 to 88.90] |

18. Secondary Outcome: Event-Free Survival (EFS) Per Kaplan-Meier Estimates
Description: EFS is defined as the time from start of treatment to the date of hematologic disease relapse/progression, graft failure, or death due to any cause. If a subject was not known to have any event, then EFS was censored at the latest date the subject was known to be alive (on or before the cut-off date).The estimated probability of event free at 1,2,6,12,18 months after start of treatment has been reported. As planned in the SAP, this outcome measure is provided for all subjects instead of per age groups.
Time Frame: 1 Month (M), 2 M, 6M, 12M, 18M
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: prob. to be event free in percentage
Arm/Group | All Subjects (Group 1, Group 2 & Group 3) | Group 4: Subjects >= 28 Days to < 2y
Number analyzed (Participants) | 45 | 0
prob. to be event free in percentage
  1 Month | 100 [100 to 100] |
  2 Months | 97.78 [88.25 to 99.68] |
  6 Months | 91.11 [78.03 to 96.57] |
  12 Months | 86.61 [72.59 to 93.75] |
  18 Months | 79.77 [64.72 to 88.93] |

19. Secondary Outcome: Failure-Free Survival (FFS)
Description: Failure-free (FF) survival was defined as the time from start date of treatment to any of the following: hematologic relapse/progression, non-relapse mortality (NRM) or addition of new systemic acute GvHD treatment. The cumulative incidence (CI) of the onset of failure event at 1,2,6,12,18,24 months after start of treatment has been reported. As planned in the SAP, this outcome measure is provided for all subjects instead of per age groups.
Time Frame: 1 Month (M), 2M, 6M, 12M, 18M, 24M
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: CI of treatment failure in percentage
Groups:
- All Subjects (Group 1, Group 2, & Group 3): All pediatric participants received ruxolitinib (RUX) regardless of dose and age group.
Arm/Group | All Subjects (Group 1, Group 2, & Group 3) | Group 4: Subjects >= 28 Days to < 2y
Number analyzed (Participants) | 45 | 0
CI of treatment failure in percentage
  1 Month | 11.11 [4.02 to 22.27] |
  2 Months | 13.33 [5.34 to 25.01] |
  6 Months | 26.67 [14.72 to 40.18] |
  12 Months | 26.67 [14.72 to 40.18] |
  18 Months | 28.97 [16.48 to 42.68] |
  24 Months | 28.97 [16.48 to 42.68] |

20. Secondary Outcome: Non Relapse Mortality (NRM)
Description: NRM is defined as the time from start of treatment to date of death not preceded by hematologic disease relapse/progression. The cumulative incidence (CI) of non-relapse mortality at 1,2,6,12,18,24 months after start of treatment has been reported. As planned in the SAP, this outcome measure is provided for all subjects instead of per age groups.
Time Frame: Month (M)1, M2, M6, M12, M18, M24
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: CI of NRM in percentage
Arm/Group | All Subjects (Group 1, Group 2 & Group 3) | Group 4: Subjects >= 28 Days to < 2y
Number analyzed (Participants) | 45 | 0
CI of NRM in percentage
  1 Month | 0.00 [NA to NA] — NA: no non-relapse mortality occurred on Month 1 |
  2 Months | 0.00 [NA to NA] — NA: no non-relapse mortality occurred on Month 2 |
  6 Months | 4.44 [0.79 to 13.47] |
  12 Months | 8.95 [2.81 to 19.58] |
  18 Months | 13.50 [5.40 to 25.31] |
  24 Months | 13.50 [5.40 to 25.31] |

21. Secondary Outcome: Incidence of Malignancy Relapse (MR)/Progression
Description: MR was defined as the time from start of treatment to hematologic malignancy relapse/progression. Calculated for patients with underlying hematologic malignant disease. The cumulative incidence (CI) of malignancy relapse/progression at 1,2,6,12,18,24 months after start of treatment has been reported. As planned in the SAP, this outcome measure is provided for all subjects instead of per age groups.
Time Frame: Month (M) 1, M2, M6, M12, M18, M24,
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: CI of MR/progression in percentage
Arm/Group | All Subjects (Group 1, Group 2 & Group 3) | Group 4: Subjects >= 28 Days to < 2y
Number analyzed (Participants) | 27 | 0
CI of MR/progression in percentage
  1 Month | 0.00 [NA to NA] — NA: no non-relapse malignancy relapse/progression occurred on Month 1 |
  2 Months | 3.70 [0.25 to 16.23] |
  6 Months | 7.41 [1.24 to 21.37] |
  12 Months | 7.41 [1.24 to 21.37] |
  18 Months | 11.28 [2.74 to 26.60] |
  24 Months | 11.28 [2.74 to 26.60] |

22. Secondary Outcome: Cumulative Incidence (CI) of cGvHD
Description: cGvHD is defined as the diagnosis of any cGvHD including mild, moderate, severe. Incidence of chronic GvHD was the time from the start of treatment to onset of chronic GvHD. Cumulative incidence of chronic GvHD was estimated, accounting for deaths without prior onset of chronic GvHD and hematologic disease relapse/progression as the competing risks. The cumulative incidence (CI) of cGvHD at 1, 2, 6, 12, 18 and 24 months after start of treatment has been reported. As planned in the SAP, this outcome measure is provided for all subjects instead of per age groups.
Time Frame: Month (M) 1, M2, M6, M12, M18, M24
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: CI of chronic GvHD in percentage
Arm/Group | All Subjects (Group 1, Group 2 & Group 3) | Group 4: Subjects >= 28 Days to < 2y
Number analyzed (Participants) | 45 | 0
CI of chronic GvHD in percentage
  1 Month | 0.00 [NA to NA] — NA: no cumulative incidence of cGvHD occurred on Month 1 |
  2 Months | 2.22 [0.17 to 10.29] |
  6 Months | 11.11 [4.01 to 22.29] |
  12 Months | 20.07 [9.80 to 32.94] |
  18 Months | 24.65 [13.11 to 38.09] |
  24 Months | 24.65 [13.11 to 38.09] |

23. Secondary Outcome: Graft Failure
Description: This was assessed by donor cell chimerism, defined as initial whole blood or marrow donor chimerism for those who had ≥5% donor cell chimerism at baseline. If donor cell chimerism declined to <5% on subsequent measurements, graft failure was declared.
Time Frame: 2 years
Population: The Efficacy Evaluable Set (EES) comprised all subjects to whom study treatment was assigned at the RP2D of ruxolitinib and who received at least one dose of study treatment at that dose level. At the end of the study there were no confirmed cases of graft failure assessment. No subjects were enrolled in Group 4.
Measure: Number; unit: Participants
Arm/Group | Group 1: Subjects ≥ 12y to < 18y - RUX 10mg BID | Group 2: Subjects ≥ 6y to < 12y - RUX 5mg BID | Group 3: Subjects ≥ 2y to < 6y - RUX 4mg/m^2 BID | Group 4: Subjects >= 28 Days to < 2y
Number analyzed (Participants) | 18 | 12 | 15 | 0
Participants | 0.0 | 0.0 | 0.0 |

24. Secondary Outcome: Questionnaire on Acceptability and Palatability
Description: Responses from the acceptability and palatability of the study drug (only for subjects administered with oral pediatric formulation starting treatment Day 1) were evaluated from a questionnaire completed by subjects, with the help from parents or caregivers as needed at the following visits: Day 1 (after first dose), Week 4 (1 month) ((after either morning or evening dose of that visit date), Week 24 (6 months) (after either morning or evening dose of that visit date). The choices for taste of the medication were, 'Very good', 'good', 'not good or bad', 'Bad', very bad. The choices for aftertaste of the medication were, 'Very good', 'Good', 'Not good or bad' , 'Bad', Very bad'. The choices for the smell of the medication were, 'Not good or bad' or 'Bad'.
Time Frame: Day 1, Week 4 (1 month), Week 24 (6 months)
Population: The Efficacy Evaluable Set (EES) comprised all subjects to whom study treatment was assigned at the RP2D of ruxolitinib and who received at least one dose of study treatment at that dose level.
Measure: Number; unit: Participants
Arm/Group | Group 2: Subjects ≥ 6y to < 12y - RUX 5mg BID Capsule | Group 3: Subjects ≥ 2y to < 6y - RUX 4mg/m^2 BID Capsule | Group 3: Subjects ≥ 2y to < 6y - RUX 4mg/m^2 BID Liquid | Group 4: Subjects >= 28 Days to < 2y
Number analyzed (Participants) | 2 | 7 | 8 | 0
Participants
  Day 1: Evaluator: Patient | 0 | 0 | 1 |
  Day 1: Evaluator: Legal guardian | 0 | 0 | 3 |
  Day 1: Evaluator: Parent | 1 | 4 | 2 |
  Day 1: Evaluator: Caregiver | 0 | 0 | 1 |
  Day 1: Evaluator: Health care professional | 1 | 3 | 1 |
  Day 1: Taste of Medicine: Very good | 0 | 0 | 3 |
  Day 1: Taste of Medicine: Good | 1 | 0 | 2 |
  Day 1: Taste of Medicine: Not good or bad | 1 | 3 | 0 |
  Day 1: Taste of Medicine: Bad | 0 | 2 | 0 |
  Day 1: Taste of Medicine: Very bad | 0 | 0 | 0 |
  Day 1: Taste of Medicine: Unable to answer the question | 0 | 2 | 3 |
  Day 1: Aftertaste of Medicine: Very good | 0 | 0 | 1 |
  Day 1: Aftertaste of Medicine: Good | 0 | 1 | 1 |
  Day 1: Aftertaste of Medicine: Not good or bad | 2 | 3 | 1 |
  Day 1: Aftertaste of Medicine: Bad | 0 | 2 | 0 |
  Day 1: Aftertaste of Medicine: Very bad | 0 | 0 | 1 |
  Day 1: Aftertaste of Medicine: Unable to answer the question | 0 | 1 | 4 |
  Day 1: Smell of Medicine: Very good | 0 | 0 | 1 |
  Day 1: Smell of Medicine: Good | 0 | 0 | 1 |
  Day 1: Smell of Medicine: Not good or bad | 2 | 4 | 3 |
  Day 1: Smell of Medicine: Bad | 0 | 1 | 0 |
  Day 1: Smell of Medicine: Very bad | 0 | 0 | 0 |
  Day 1: Smell of Medicine: Unable to answer the question | 0 | 2 | 3 |
  Week 4: Evaluatohr: Legal guardian: number analyzed (Participants) | 2 | 6 | 8 | 0
  Week 4: Evaluatohr: Legal guardian | 0 | 1 | 2 |
  Week 4: Evaluator: Parent: number analyzed (Participants) | 2 | 6 | 8 | 0
  Week 4: Evaluator: Parent | 1 | 5 | 4 |
  Week 4: Evaluator: Health care professional: number analyzed (Participants) | 2 | 6 | 8 | 0
  Week 4: Evaluator: Health care professional | 1 | 0 | 2 |
  Week 4: Taste of Medicine: Very good: number analyzed (Participants) | 2 | 6 | 8 | 0
  Week 4: Taste of Medicine: Very good | 0 | 0 | 0 |
  Week 4: Taste of Medicine: Good: number analyzed (Participants) | 2 | 6 | 8 | 0
  Week 4: Taste of Medicine: Good | 2 | 1 | 4 |
  Week 4: Taste of Medicine: Not good or bad: number analyzed (Participants) | 2 | 6 | 8 | 0
  Week 4: Taste of Medicine: Not good or bad | 0 | 4 | 1 |
  Week 4: Taste of Medicine: Bad: number analyzed (Participants) | 2 | 6 | 8 | 0
  Week 4: Taste of Medicine: Bad | 0 | 0 | 0 |
  Week 4: Taste of Medicine: Very bad: number analyzed (Participants) | 2 | 6 | 8 | 0
  Week 4: Taste of Medicine: Very bad | 0 | 1 | 0 |
  Week 4: Taste of Medicine: Unable to answer the question: number analyzed (Participants) | 2 | 6 | 8 | 0
  Week 4: Taste of Medicine: Unable to answer the question | 0 | 0 | 3 |
  Week 4: Aftertaste of Medicine: Very good: number analyzed (Participants) | 2 | 6 | 8 | 0
  Week 4: Aftertaste of Medicine: Very good | 0 | 0 | 0 |
  Week 4: Aftertaste of Medicine: Good: number analyzed (Participants) | 2 | 6 | 8 | 0
  Week 4: Aftertaste of Medicine: Good | 0 | 1 | 2 |
  Week 4: Aftertaste of Medicine: Not good or bad: number analyzed (Participants) | 2 | 6 | 8 | 0
  Week 4: Aftertaste of Medicine: Not good or bad | 2 | 3 | 1 |
  Week 4: Aftertaste of Medicine: Bad: number analyzed (Participants) | 2 | 6 | 8 | 0
  Week 4: Aftertaste of Medicine: Bad | 0 | 1 | 0 |
  Week 4: Aftertaste of Medicine: Very bad: number analyzed (Participants) | 2 | 6 | 8 | 0
  Week 4: Aftertaste of Medicine: Very bad | 0 | 0 | 0 |
  Week 4: Aftertaste of Medicine: Unable to answer the question: number analyzed (Participants) | 2 | 6 | 8 | 0
  Week 4: Aftertaste of Medicine: Unable to answer the question | 0 | 1 | 5 |
  Week 4: Smell of Medicine: Very good: number analyzed (Participants) | 2 | 6 | 8 | 0
  Week 4: Smell of Medicine: Very good | 0 | 0 | 1 |
  Week 4: Smell of Medicine: Good: number analyzed (Participants) | 2 | 6 | 8 | 0
  Week 4: Smell of Medicine: Good | 0 | 0 | 0 |
  Week 4: Smell of Medicine: Not good or bad: number analyzed (Participants) | 2 | 6 | 8 | 0
  Week 4: Smell of Medicine: Not good or bad | 2 | 5 | 3 |
  Week 4: Smell of Medicine: Bad: number analyzed (Participants) | 2 | 6 | 8 | 0
  Week 4: Smell of Medicine: Bad | 0 | 0 | 1 |
  Week 4: Smell of Medicine: Very bad: number analyzed (Participants) | 2 | 6 | 8 | 0
  Week 4: Smell of Medicine: Very bad | 0 | 0 | 0 |
  Week 4: Smell of Medicine: Unable to answer the question: number analyzed (Participants) | 2 | 6 | 8 | 0
  Week 4: Smell of Medicine: Unable to answer the question | 0 | 1 | 3 |
  Week 24: Evaluator: Patient: number analyzed (Participants) | 0 | 2 | 2 | 0
  Week 24: Evaluator: Patient |  | 1 | 1 |
  Week 24: Evaluator: Parent: number analyzed (Participants) | 0 | 2 | 2 | 0
  Week 24: Evaluator: Parent |  | 1 | 0 |
  Week 24: Evaluator: Health care professional: number analyzed (Participants) | 0 | 2 | 2 | 0
  Week 24: Evaluator: Health care professional |  | 0 | 1 |
  Week 24: Taste of Medicine: Very good: number analyzed (Participants) | 0 | 2 | 2 | 0
  Week 24: Taste of Medicine: Very good |  | 0 | 2 |
  Week 24: Taste of Medicine: Good: number analyzed (Participants) | 0 | 2 | 2 | 0
  Week 24: Taste of Medicine: Good |  | 1 | 0 |
  Week 24: Taste of Medicine: Not good or bad: number analyzed (Participants) | 0 | 2 | 2 | 0
  Week 24: Taste of Medicine: Not good or bad |  | 1 | 0 |
  Week 24: Taste of Medicine: Bad: number analyzed (Participants) | 0 | 2 | 2 | 0
  Week 24: Taste of Medicine: Bad |  | 0 | 0 |
  Week 24: Taste of Medicine: Very bad: number analyzed (Participants) | 0 | 2 | 2 | 0
  Week 24: Taste of Medicine: Very bad |  | 0 | 0 |
  Week 24: Taste of Medicine: Unable to answer the question: number analyzed (Participants) | 0 | 2 | 2 | 0
  Week 24: Taste of Medicine: Unable to answer the question |  | 0 | 0 |
  Week 24: Aftertaste of Medicine: Very good: number analyzed (Participants) | 0 | 2 | 2 | 0
  Week 24: Aftertaste of Medicine: Very good |  | 0 | 1 |
  Week 24: Aftertaste of Medicine: Not good or bad: number analyzed (Participants) | 0 | 2 | 2 | 0
  Week 24: Aftertaste of Medicine: Not good or bad |  | 2 | 0 |
  Week 24: Aftertaste of Medicine: Unable to answer the question: number analyzed (Participants) | 0 | 2 | 2 | 0
  Week 24: Aftertaste of Medicine: Unable to answer the question |  | 0 | 1 |
  Week 24: Smell of Medicine: Very good: number analyzed (Participants) | 0 | 2 | 2 | 0
  Week 24: Smell of Medicine: Very good |  | 0 | 1 |
  Week 24: Smell of Medicine: Good: number analyzed (Participants) | 0 | 2 | 2 | 0
  Week 24: Smell of Medicine: Good |  | 0 | 1 |
  Week 24: Smell of Medicine: Not good or bad: number analyzed (Participants) | 0 | 2 | 2 | 0
  Week 24: Smell of Medicine: Not good or bad |  | 2 | 0 |
  Week 24: Smell of Medicine: Bad: number analyzed (Participants) | 0 | 2 | 2 | 0
  Week 24: Smell of Medicine: Bad |  | 0 | 0 |
  Week 24: Smell of Medicine: Very bad: number analyzed (Participants) | 0 | 2 | 2 | 0
  Week 24: Smell of Medicine: Very bad |  | 0 | 0 |
  Week 24: Smell of Medicine: Unable to answer the question: number analyzed (Participants) | 0 | 2 | 2 | 0
  Week 24: Smell of Medicine: Unable to answer the question |  | 0 | 0 |

25. Secondary Outcome: PK Parameter - Maximum Serum Concentration (Cmax) Versus Efficacy
Description: To assess pharmacokinetic/pharmacodynamic relationship (comparison of Cmax with efficacy). Cmax: The maximum (peak) observed plasma drug concentration.
Time Frame: 24 weeks
Population: Based on PK-safety/PK-efficacy analyses conducted in adult acute & chronic GvHD studies (REACH2 & REACH3), AUC was considered the most informative PK metric to assess the relationship between PK (exposure to ruxolitinib) and efficacy/safety/pharmadynamic (PD) parameters. Thus, to assess PK-safety, PK-efficacy and PK-PD biomarker in pediatric GvHD patients, AUC was selected as the PK measure of interest; the relationship between Cmax/Ctrough and efficacy/safety/PD biomarker was not investigated.
Arm/Group | Group 1: Subjects ≥ 12y to < 18y - RUX 10mg BID Tablet | Group 2: Subjects ≥ 6y to < 12y - RUX 5mg BID Tablet | Group 2: Subjects ≥ 6y to < 12y - RUX 5mg BID Capsule | Group 3: Subjects ≥ 2y to < 6y - RUX 4mg/m^2 BID Capsule | Group 3: Subjects ≥ 2y to < 6y - RUX 4mg/m^2 BID Liquid | Group 4: Subjects >= 28 Days to < 2y
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

26. Secondary Outcome: PK Parameter: Minimum Serum Concentration (Ctrough) Versus Safety
Description: To assess pharmacokinetic/pharmacodynamic relationships (comparison of Ctrough with safety). Ctrough: The minimum observed plasma concentration at the end of an administration interval (corresponding to the pre-dose concentration prior to the following administration).
Time Frame: 24 weeks
Population: as for outcome 25
Arm/Group | Group 1: Subjects ≥ 12y to < 18y - RUX 10mg BID Tablet | Group 2: Subjects ≥ 6y to < 12y - RUX 5mg BID Tablet | Group 2: Subjects ≥ 6y to < 12y - RUX 5mg BID Capsule | Group 3: Subjects ≥ 2y to < 6y - RUX 4mg/m^2 BID Capsule | Group 3: Subjects ≥ 2y to < 6y - RUX 4mg/m^2 BID Liquid | Group 4: Subjects >= 28 Days to < 2y
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

27. Secondary Outcome: PK Parameter: Cmax Versus Safety
Description: To assess pharmacokinetic/pharmacodynamics relationship (comparison of Cmax with safety). Cmax: The maximum (peak) observed plasma drug concentration.
Time Frame: 24 weeks
Population: as for outcome 25
Arm/Group | Group 1: Subjects ≥ 12y to < 18y - RUX 10mg BID Tablet | Group 2: Subjects ≥ 6y to < 12y - RUX 5mg BID Tablet | Group 2: Subjects ≥ 6y to < 12y - RUX 5mg BID Capsule | Group 3: Subjects ≥ 2y to < 6y - RUX 4mg/m^2 BID Capsule | Group 3: Subjects ≥ 2y to < 6y - RUX 4mg/m^2 BID Liquid | Group 4: Subjects >= 28 Days to < 2y
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

28. Secondary Outcome: PK Parameter: Ctrough Versus Efficacy
Description: To assess pharmacokinetic/pharmacodynamics relationship (comparison of Ctrough with efficacy). Ctrough: The minimum observed plasma concentration at the end of an administration interval (corresponding to the pre-dose concentration prior to the following administration).
Time Frame: 24 weeks
Population: as for outcome 25
Arm/Group | Group 1: Subjects ≥ 12y to < 18y - RUX 10mg BID Tablet | Group 2: Subjects ≥ 6y to < 12y - RUX 5mg BID Tablet | Group 2: Subjects ≥ 6y to < 12y - RUX 5mg BID Capsule | Group 3: Subjects ≥ 2y to < 6y - RUX 4mg/m^2 BID Capsule | Group 3: Subjects ≥ 2y to < 6y - RUX 4mg/m^2 BID Liquid | Group 4: Subjects >= 28 Days to < 2y
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

29. Secondary Outcome: PK Parameter: Profile of Biomarker Concentration Changes Across Different AUC Quantile Groups
Description: Describe the relationship between AUC and PD biomarkers. Provide profile of biomarker concentration changes across different AUC quantile groups from baseline. This analysis includes subjects from F12201 study. Population was divided by four level of exposure using AUClast Day 1 quartiles. As planned in SAP, this outcome measure is provided for all subjects instead of per age groups.
Time Frame: Week 4
Population: PAS included all subjects (subjs) who provided at least 1 evaluable PK concentration. For a concentration to be evaluable, subjs were required to: Take the dose of ruxolitinib prior to PK sample; For pre-dose samples, to not vomit within 2 hrs after the previous dosing of ruxolitinib prior to sampling; for post-dose samples, to not vomit within 2 hrs after the dosing of ruxolitinib. Subjs in each age grp were combined as pre-specified in the Stats Analysis Plan. No subjs were enrolled in Grp 4.
Measure: Median (Inter-Quartile Range); unit: Week 4 percentage change from baseline
Groups:
- AUClast Day 1: 1st Quartile; AUClast Day 1: 2nd Quartile; AUClast Day 1: 3rd Quartile; AUClast Day 1: 4th Quartile: AUClast: The AUC from time zero to the last measurable concentration sampling time (Tlast).
Arm/Group | AUClast Day 1: 1st Quartile | AUClast Day 1: 2nd Quartile | AUClast Day 1: 3rd Quartile | AUClast Day 1: 4th Quartile | Group 4: Subjects >= 28 Days to < 2y
Number analyzed (Participants) | 7 | 8 | 7 | 8 | 0
Week 4 percentage change from baseline
  Biomarker: IL10 | 0.00 [-85.64 to 225.33] | -22.43 [-76.22 to 0.00] | -79.71 [-89.63 to -47.49] | -50.72 [-58.01 to 73.55] |
  Biomarker: IL6 | -59.48 [-69.78 to 0.00] | -10.40 [-80.48 to 0.00] | 0.00 [-67.78 to 0.00] | 181.48 [0.00 to 376.54] |
  Biomarker: IL8 | -63.63 [-70.48 to -21.03] | 42.57 [-22.15 to 201.65] | 31.79 [-48.56 to 329.67] | 60.02 [-41.74 to 280.49] |
  Biomarker: TNFA | -61.45 [-74.05 to -56.96] | 0.00 [-31.03 to 33.67] | -35.34 [-65.90 to -1.41] | 21.49 [-48.52 to 311.76] |
  Biomarker: CD4 Assay (CD4 T cells) (%), | -40.49 [-42.67 to -35.51] | 98.07 [16.40 to 206.34] | -3.07 [-17.66 to 115.79] | -42.67 [-62.47 to 92.71] |
  Biomarker: CD8 Assay (CD8 T cells) (%), | -51.80 [-69.95 to -20.07] | 64.71 [6.18 to 118.32] | 104.17 [-34.38 to 270.84] | 33.77 [-76.27 to 114.61] |
  Biomarker: FOXP3 Assay (Treg cells) (%) | 115.79 [-26.03 to 124.24] | 43.15 [2.08 to 52.17] | 57.14 [-16.49 to 79.73] | -11.11 [-60.56 to 119.05] |
  Biomarker: IL14A Assay (Th17 cells) (%) | 5.33 [-33.75 to 10.78] | 140.91 [-25.53 to 570.83] | -7.69 [-18.92 to 131.25] | 38.73 [-57.47 to 203.45] |
  Biomarker: LRP5 Assay (B cells) (%), | -15.00 [-30.00 to 122.78] | 25.78 [-42.86 to 300.00] | 140.00 [37.80 to 142.86] | 105.26 [-30.77 to 650.00] |
  MVD Assay (NK cells) (%) | -23.82 [-24.21 to 65.52] | 61.81 [34.74 to 98.53] | 22.54 [-18.99 to 69.08] | -0.71 [-34.19 to 72.62] |

30. Secondary Outcome: PK Parameter: Cmax Versus PD Biomarkers
Description: To assess pharmacokinetic/pharmacodynamic relationship (comparison of Cmax with PD biomarkers). Cmax: The maximum (peak) observed plasma drug concentration.
Time Frame: 24 weeks
Population: as for outcome 25
Arm/Group | Group 1: Subjects ≥ 12y to < 18y - RUX 10mg BID | Group 2: Subjects ≥ 6y to < 12y - RUX 5mg BID | Group 2: Subjects ≥ 6y to < 12y - RUX 5mg BID Capsule | Group 3: Subjects ≥ 2y to < 6y - RUX 4mg/m^2 BID Capsule | Group 3: Subjects ≥ 2y to < 6y - RUX 4mg/m^2 BID Liquid | Group 4: Subjects >= 28 Days to < 2y
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

31. Secondary Outcome: PK Parameter: Ctrough Versus PD Biomarkers
Description: To assess pharmacokinetic/pharmacodynamics relationship (Ctrough with PD biomarkers). Ctrough: The minimum observed plasma concentration at the end of an administration interval (corresponding to the pre-dose concentration prior to the following administration).
Time Frame: 24 weeks
Population: as for outcome 25
Arm/Group | Group 1: Subjects ≥ 12y to < 18y - RUX 10mg BID | Group 2: Subjects ≥ 6y to < 12y - RUX 5mg BID | Group 2: Subjects ≥ 6y to < 12y - RUX 5mg BID Capsule | Group 3: Subjects ≥ 2y to < 6y - RUX 4mg/m^2 BID Capsule | Group 3: Subjects ≥ 2y to < 6y - RUX 4mg/m^2 BID Liquid | Group 4: Subjects >= 28 Days to < 2y
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

32. Secondary Outcome: Percentage of Patients Who Achieved Best Overall Response (BOR) up to Day 28
Description: The best overall response (BOR) was defined as percentage of participants with (complete response (CR) or partial response (PR) at any time point and up to and including Day 28 and before the start of additional systemic therapy for acute GvHD (aGvHD).
Time Frame: Up to 28 days and before start of additional aGvHD therapy
Population: as for outcome 9
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Groups:
- Group 1: ≥ 12y to < 18y - RUX 10mg BID: All patients received ruxolitinib (RUX) 10 mg BID.
Arm/Group | Group 1: ≥ 12y to < 18y - RUX 10mg BID | Group 2: Subjects ≥ 6y to < 12y - RUX 5mg BID | Group 3: Subjects ≥ 2y to < 6y - RUX 4mg/m^2 BID | Group 4: Subjects >= 28 Days to < 2y
Number analyzed (Participants) | 18 | 12 | 15 | 0
Percentage of participants | 94.4 [76.2 to 99.7] | 91.7 [66.1 to 99.6] | 93.3 [72.1 to 99.7] |

33. Post Hoc Outcome: All Collected Deaths
Description: Adverse events and on-treatment deaths were collected from the first dose of study treatment up to 30 days after last dose of study medication, for a maximum duration of 380 days.
  Post-treatment survival follow-up deaths were collected 31 days after last dose of study medication until the end of the study, up to approx. 23 months.
Time Frame: AEs & On-treatment deaths: Up to approx. 380 days (13 months), Post-treatment survival follow-up deaths: Up to approx. 23 months after the end of treatment
Population: Clinical database population: all treated patients, patients who died during screening and patients who were enrolled into the study. No subjects were enrolled in Group 4.
Measure: Number; unit: Participants
Arm/Group | Group 1: Subjects ≥ 12y to < 18y - RUX 10mg BID | Group 2: Subjects ≥ 6y to < 12y - RUX 5mg BID | Group 3: Subjects ≥ 2y to < 6y - RUX 4mg/m^2 BID | Group 4: Subjects >= 28 Days to < 2y
Number analyzed (Participants) | 18 | 12 | 15 | 0
Participants
  Total deaths | 6 | 2 | 1 |
  On-treatment deaths | 0 | 0 | 0 |
  Post-treatment deaths | 6 | 2 | 1 |

ADVERSE EVENTS:
Time Frame: Adverse events and on-treatment deaths were collected from the first dose of study treatment up to 30 days after last dose of study medication, for a maximum duration of 380 days. Post-treatment survival follow-up deaths were collected 31 days after last dose of study medication until the end of the study, up to approx. 23 months.
Description: Any sign or symptom that occurs during the conduct of the trial and safety follow-up. Deaths in the post treatment survival follow-up are not considered Adverse Events. The total number at risk in the post treatment survival includes patients that entered the post treatment survival follow-up period. No subjects were enrolled in Group 4.
Groups:
- Group 1: Subjects >=12y - <18y - RUX 10mg (On-treatment); Group 2: Subjects >=6y - <12y - RUX 5mg (On-treatment); Group 3: Subjects >=2y - <6y - RUX 4mg/m2 (On-treatment): On-treatment period: from first dose of study treatment up to 30 days post-treatment
- All Subjects: All subjects from Group 1, Group 2 and Group 3 who were enrolled and participated in the study
- Group 1: Subjects ≥ 12y to < 18y - RUX 10mg (Post-treatment Survival Follow-up); Group 2: Subjects ≥ 6y to < 12y - RUX 5mg (Post-treatment Survival Follow-up); Group 3: Subjects ≥ 2y to < 6y - RUX 4mg/m2 (Post-treatment Survival Follow-up): Deaths collected in the post- treatment survival follow-up phase (starting from day 31 post- treatment). No AEs were collected during this period
Arm/Group | Group 1: Subjects >=12y - <18y - RUX 10mg (On-treatment) | Group 2: Subjects >=6y - <12y - RUX 5mg (On-treatment) | Group 3: Subjects >=2y - <6y - RUX 4mg/m2 (On-treatment) | All Subjects | Group 1: Subjects ≥ 12y to < 18y - RUX 10mg (Post-treatment Survival Follow-up) | Group 2: Subjects ≥ 6y to < 12y - RUX 5mg (Post-treatment Survival Follow-up) | Group 3: Subjects ≥ 2y to < 6y - RUX 4mg/m2 (Post-treatment Survival Follow-up) | Group 4: Subjects >= 28 Days to < 2y
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/12 | 0/15 | 0/45 | 6/18 | 2/12 | 1/15 | 0/0
Serious Adverse Events (participants affected / at risk) | 11/18 | 7/12 | 6/15 | 24/45 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 18/18 | 12/12 | 15/15 | 45/45 | 0/0 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: Subjects >=12y - <18y - RUX 10mg (On-treatment) (N=18) | Group 2: Subjects >=6y - <12y - RUX 5mg (On-treatment) (N=12) | Group 3: Subjects >=2y - <6y - RUX 4mg/m2 (On-treatment) (N=15) | All Subjects (N=45) | Group 1: Subjects ≥ 12y to < 18y - RUX 10mg (Post-treatment Survival Follow-up) (N=0) | Group 2: Subjects ≥ 6y to < 12y - RUX 5mg (Post-treatment Survival Follow-up) (N=0) | Group 3: Subjects ≥ 2y to < 6y - RUX 4mg/m2 (Post-treatment Survival Follow-up) (N=0) | Group 4: Subjects >= 28 Days to < 2y (N=0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 2 | NA | NA | NA | NA
Haemorrhagic disorder (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Immune thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0 | 1 | NA | NA | NA | NA
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Intestinal perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | NA | NA | NA | NA
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | NA | NA | NA | NA
Pyrexia (General disorders) | 1 | 1 | 2 | 4 | NA | NA | NA | NA
Graft versus host disease in gastrointestinal tract (Immune system disorders) | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Adenovirus infection (Infections and infestations) | 0 | 1 | 0 | 1 | NA | NA | NA | NA
COVID-19 (Infections and infestations) | 0 | 0 | 1 | 1 | NA | NA | NA | NA
Cytomegalovirus viraemia (Infections and infestations) | 0 | 0 | 1 | 1 | NA | NA | NA | NA
Device related infection (Infections and infestations) | 0 | 1 | 0 | 1 | NA | NA | NA | NA
Eye infection viral (Infections and infestations) | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 1 | NA | NA | NA | NA
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Sepsis (Infections and infestations) | 0 | 1 | 1 | 2 | NA | NA | NA | NA
Septic shock (Infections and infestations) | 2 | 0 | 0 | 2 | NA | NA | NA | NA
Skin infection (Infections and infestations) | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Viral haemorrhagic cystitis (Infections and infestations) | 1 | 0 | 1 | 2 | NA | NA | NA | NA
Transplant dysfunction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Adenovirus test positive (Investigations) | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Cytomegalovirus test positive (Investigations) | 0 | 0 | 1 | 1 | NA | NA | NA | NA
Neutrophil count decreased (Investigations) | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Platelet count decreased (Investigations) | 1 | 0 | 0 | 1 | NA | NA | NA | NA
White blood cell count decreased (Investigations) | 0 | 1 | 0 | 1 | NA | NA | NA | NA
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | NA | NA | NA | NA
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 | 0 | 1 | 1 | NA | NA | NA | NA
Acute kidney injury (Renal and urinary disorders) | 2 | 0 | 0 | 2 | NA | NA | NA | NA
Renal failure (Renal and urinary disorders) | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Shock haemorrhagic (Vascular disorders) | 0 | 1 | 0 | 1 | NA | NA | NA | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: Subjects >=12y - <18y - RUX 10mg (On-treatment) (N=18) | Group 2: Subjects >=6y - <12y - RUX 5mg (On-treatment) (N=12) | Group 3: Subjects >=2y - <6y - RUX 4mg/m2 (On-treatment) (N=15) | All Subjects (N=45) | Group 1: Subjects ≥ 12y to < 18y - RUX 10mg (Post-treatment Survival Follow-up) (N=0) | Group 2: Subjects ≥ 6y to < 12y - RUX 5mg (Post-treatment Survival Follow-up) (N=0) | Group 3: Subjects ≥ 2y to < 6y - RUX 4mg/m2 (Post-treatment Survival Follow-up) (N=0) | Group 4: Subjects >= 28 Days to < 2y (N=0)
Anaemia (Blood and lymphatic system disorders) | 6 | 5 | 9 | 20 | NA | NA | NA | NA
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 2 | NA | NA | NA | NA
Hyperleukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | NA | NA | NA | NA
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | NA | NA | NA | NA
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Leukopenia (Blood and lymphatic system disorders) | 3 | 0 | 0 | 3 | NA | NA | NA | NA
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Neutropenia (Blood and lymphatic system disorders) | 6 | 2 | 1 | 9 | NA | NA | NA | NA
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 0 | 2 | 8 | NA | NA | NA | NA
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Bradycardia (Cardiac disorders) | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Cardiac failure (Cardiac disorders) | 0 | 1 | 0 | 1 | NA | NA | NA | NA
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 1 | NA | NA | NA | NA
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 1 | NA | NA | NA | NA
Ventricular fibrillation (Cardiac disorders) | 0 | 1 | 0 | 1 | NA | NA | NA | NA
Adrenal insufficiency (Endocrine disorders) | 1 | 2 | 1 | 4 | NA | NA | NA | NA
Cushingoid (Endocrine disorders) | 1 | 1 | 0 | 2 | NA | NA | NA | NA
Secondary adrenocortical insufficiency (Endocrine disorders) | 0 | 0 | 1 | 1 | NA | NA | NA | NA
Dry eye (Eye disorders) | 1 | 0 | 1 | 2 | NA | NA | NA | NA
Eye disorder (Eye disorders) | 0 | 1 | 0 | 1 | NA | NA | NA | NA
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 3 | 5 | NA | NA | NA | NA
Anal fissure (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Angular cheilitis (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Constipation (Gastrointestinal disorders) | 1 | 2 | 2 | 5 | NA | NA | NA | NA
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 1 | 5 | NA | NA | NA | NA
Intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | NA | NA | NA | NA
Vomiting (Gastrointestinal disorders) | 1 | 1 | 2 | 4 | NA | NA | NA | NA
Asthenia (General disorders) | 0 | 1 | 0 | 1 | NA | NA | NA | NA
Catheter site erythema (General disorders) | 0 | 1 | 0 | 1 | NA | NA | NA | NA
Chills (General disorders) | 0 | 1 | 0 | 1 | NA | NA | NA | NA
Face oedema (General disorders) | 0 | 1 | 0 | 1 | NA | NA | NA | NA
Oedema (General disorders) | 0 | 0 | 1 | 1 | NA | NA | NA | NA
Oedema peripheral (General disorders) | 0 | 1 | 0 | 1 | NA | NA | NA | NA
Pyrexia (General disorders) | 2 | 2 | 2 | 6 | NA | NA | NA | NA
Hepatic steatosis (Hepatobiliary disorders) | 0 | 1 | 0 | 1 | NA | NA | NA | NA
Hepatotoxicity (Hepatobiliary disorders) | 2 | 0 | 0 | 2 | NA | NA | NA | NA
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Acute graft versus host disease in intestine (Immune system disorders) | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Allergy to immunoglobulin therapy (Immune system disorders) | 0 | 0 | 1 | 1 | NA | NA | NA | NA
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 1 | NA | NA | NA | NA
Graft versus host disease in skin (Immune system disorders) | 0 | 1 | 0 | 1 | NA | NA | NA | NA
Hypogammaglobulinaemia (Immune system disorders) | 1 | 0 | 1 | 2 | NA | NA | NA | NA
Atypical pneumonia (Infections and infestations) | 0 | 0 | 1 | 1 | NA | NA | NA | NA
Bacteraemia (Infections and infestations) | 0 | 1 | 0 | 1 | NA | NA | NA | NA
Bronchitis (Infections and infestations) | 2 | 0 | 1 | 3 | NA | NA | NA | NA
COVID-19 (Infections and infestations) | 0 | 0 | 2 | 2 | NA | NA | NA | NA
Cystitis (Infections and infestations) | 2 | 0 | 0 | 2 | NA | NA | NA | NA
Cytomegalovirus infection (Infections and infestations) | 3 | 0 | 0 | 3 | NA | NA | NA | NA
Cytomegalovirus infection reactivation (Infections and infestations) | 2 | 1 | 1 | 4 | NA | NA | NA | NA
Cytomegalovirus viraemia (Infections and infestations) | 0 | 0 | 1 | 1 | NA | NA | NA | NA
Device related infection (Infections and infestations) | 1 | 0 | 1 | 2 | NA | NA | NA | NA
Ear infection (Infections and infestations) | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Epstein-Barr virus infection (Infections and infestations) | 1 | 0 | 1 | 2 | NA | NA | NA | NA
Epstein-Barr virus infection reactivation (Infections and infestations) | 0 | 1 | 3 | 4 | NA | NA | NA | NA
Fungal foot infection (Infections and infestations) | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Fungal infection (Infections and infestations) | 0 | 0 | 1 | 1 | NA | NA | NA | NA
Herpes simplex (Infections and infestations) | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Klebsiella infection (Infections and infestations) | 0 | 1 | 0 | 1 | NA | NA | NA | NA
Mucosal infection (Infections and infestations) | 2 | 0 | 0 | 2 | NA | NA | NA | NA
Nail infection (Infections and infestations) | 0 | 0 | 1 | 1 | NA | NA | NA | NA
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 1 | NA | NA | NA | NA
Oral candidiasis (Infections and infestations) | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Oral herpes (Infections and infestations) | 0 | 1 | 0 | 1 | NA | NA | NA | NA
Otitis externa (Infections and infestations) | 0 | 1 | 0 | 1 | NA | NA | NA | NA
Otitis media (Infections and infestations) | 0 | 0 | 1 | 1 | NA | NA | NA | NA
Rhinitis (Infections and infestations) | 1 | 0 | 1 | 2 | NA | NA | NA | NA
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 1 | NA | NA | NA | NA
Staphylococcal sepsis (Infections and infestations) | 0 | 1 | 0 | 1 | NA | NA | NA | NA
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Urinary tract infection (Infections and infestations) | 0 | 1 | 1 | 2 | NA | NA | NA | NA
Varicella zoster virus infection (Infections and infestations) | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Viraemia (Infections and infestations) | 0 | 1 | 0 | 1 | NA | NA | NA | NA
Viral haemorrhagic cystitis (Infections and infestations) | 0 | 0 | 1 | 1 | NA | NA | NA | NA
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 1 | 1 | NA | NA | NA | NA
Vulvovaginitis (Infections and infestations) | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Anaphylactic transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | NA | NA | NA | NA
Post procedural contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | NA | NA | NA | NA
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | NA | NA | NA | NA
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | NA | NA | NA | NA
Adenovirus test positive (Investigations) | 0 | 0 | 2 | 2 | NA | NA | NA | NA
Alanine aminotransferase increased (Investigations) | 5 | 2 | 2 | 9 | NA | NA | NA | NA
Amylase increased (Investigations) | 0 | 1 | 0 | 1 | NA | NA | NA | NA
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 2 | 3 | NA | NA | NA | NA
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Blood cholesterol increased (Investigations) | 1 | 0 | 1 | 2 | NA | NA | NA | NA
Blood creatinine increased (Investigations) | 1 | 1 | 2 | 4 | NA | NA | NA | NA
C-reactive protein increased (Investigations) | 0 | 1 | 0 | 1 | NA | NA | NA | NA
Cytomegalovirus test positive (Investigations) | 1 | 1 | 4 | 6 | NA | NA | NA | NA
Epstein-Barr virus test positive (Investigations) | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Gamma-glutamyltransferase increased (Investigations) | 1 | 2 | 2 | 5 | NA | NA | NA | NA
Lipase increased (Investigations) | 2 | 0 | 1 | 3 | NA | NA | NA | NA
Lymphocyte count decreased (Investigations) | 1 | 1 | 1 | 3 | NA | NA | NA | NA
Neutrophil count decreased (Investigations) | 5 | 2 | 5 | 12 | NA | NA | NA | NA
Platelet count decreased (Investigations) | 0 | 2 | 6 | 8 | NA | NA | NA | NA
Prothrombin time abnormal (Investigations) | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Roseolovirus test positive (Investigations) | 0 | 0 | 1 | 1 | NA | NA | NA | NA
SARS-CoV-2 test negative (Investigations) | 0 | 1 | 0 | 1 | NA | NA | NA | NA
Transaminases increased (Investigations) | 2 | 0 | 0 | 2 | NA | NA | NA | NA
Weight decreased (Investigations) | 0 | 2 | 0 | 2 | NA | NA | NA | NA
Weight increased (Investigations) | 1 | 2 | 0 | 3 | NA | NA | NA | NA
White blood cell count decreased (Investigations) | 0 | 2 | 5 | 7 | NA | NA | NA | NA
Central obesity (Metabolism and nutrition disorders) | 1 | 1 | 1 | 3 | NA | NA | NA | NA
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | NA | NA | NA | NA
Folate deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | NA | NA | NA | NA
Hyperferritinaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | NA | NA | NA | NA
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 0 | 0 | 3 | NA | NA | NA | NA
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | NA | NA | NA | NA
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 2 | NA | NA | NA | NA
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 3 | 0 | 5 | NA | NA | NA | NA
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | NA | NA | NA | NA
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 3 | 0 | 7 | NA | NA | NA | NA
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 3 | NA | NA | NA | NA
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 3 | NA | NA | NA | NA
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Amyotrophy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | NA | NA | NA | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | NA | NA | NA | NA
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | NA | NA | NA | NA
Muscle contracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2 | NA | NA | NA | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2 | NA | NA | NA | NA
Generalised tonic-clonic seizure (Nervous system disorders) | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Headache (Nervous system disorders) | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Neuralgia (Nervous system disorders) | 0 | 1 | 0 | 1 | NA | NA | NA | NA
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 1 | NA | NA | NA | NA
Post herpetic neuralgia (Nervous system disorders) | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 | 1 | 0 | 1 | NA | NA | NA | NA
Restless legs syndrome (Nervous system disorders) | 0 | 1 | 0 | 1 | NA | NA | NA | NA
Depression (Psychiatric disorders) | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 1 | NA | NA | NA | NA
Cystitis haemorrhagic (Renal and urinary disorders) | 2 | 1 | 0 | 3 | NA | NA | NA | NA
Glycosuria (Renal and urinary disorders) | 0 | 0 | 1 | 1 | NA | NA | NA | NA
Ketonuria (Renal and urinary disorders) | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Micturition urgency (Renal and urinary disorders) | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Polyuria (Renal and urinary disorders) | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Proteinuria (Renal and urinary disorders) | 2 | 1 | 1 | 4 | NA | NA | NA | NA
Renal impairment (Renal and urinary disorders) | 0 | 1 | 0 | 1 | NA | NA | NA | NA
Urinary tract pain (Renal and urinary disorders) | 0 | 0 | 1 | 1 | NA | NA | NA | NA
Penile erosion (Reproductive system and breast disorders) | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Bronchial disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | NA | NA | NA | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 3 | NA | NA | NA | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | NA | NA | NA | NA
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 2 | NA | NA | NA | NA
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | NA | NA | NA | NA
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | NA | NA | NA | NA
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2 | NA | NA | NA | NA
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | NA | NA | NA | NA
Bullous haemorrhagic dermatosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | NA | NA | NA | NA
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | NA | NA | NA | NA
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 3 | NA | NA | NA | NA
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 2 | NA | NA | NA | NA
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | NA | NA | NA | NA
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | NA | NA | NA | NA
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 2 | NA | NA | NA | NA
Hirsutism (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 2 | NA | NA | NA | NA
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | NA | NA | NA | NA
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | NA | NA | NA | NA
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | NA | NA | NA | NA
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 2 | NA | NA | NA | NA
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 3 | NA | NA | NA | NA
Skin fissures (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Skin striae (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Capillary leak syndrome (Vascular disorders) | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Hypertension (Vascular disorders) | 2 | 2 | 5 | 9 | NA | NA | NA | NA
Microangiopathy (Vascular disorders) | 1 | 0 | 0 | 1 | NA | NA | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Study Protocol (2022-06-24): https://cdn.clinicaltrials.gov/large-docs/15/NCT03491215/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-10): https://cdn.clinicaltrials.gov/large-docs/15/NCT03491215/SAP_001.pdf